CLINICAL TRIAL: NCT07230067
Title: The Impact of Platelet Transfusion Therapy on 28-day Mortality in Septic Patients With Thrombocytopenia During ICU Stay: a Multicenter Retrospective Observational Study
Brief Title: Sepsis-associated Thrombocytopenia and Platelet Transfusion （STAPT）
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-392
Record Dates: First submitted 2025-08-29; First posted 2025-11-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Sepsis and Coagulopathy
Keywords: Sepsis-Associated Thrombocytopenia; Platelet infusion; mortality; sepsis; platelet
MeSH Terms: conditions — Sepsis; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Platelet Transfusion Group: Platelet Transfusion within 14 days after ICU admission
  Interventions: Other: SAT patients
- No Platelet Transfusion Group: No Platelet Transfusion within 14 days after ICU admission
  Interventions: Other: SAT patients

INTERVENTIONS:
Other: SAT patients — Whether or not the SAT patients received Platelet infusion

SUMMARY:
Currently, there are no multicenter studies on platelet transfusion for SAT patients, and the benefits and risks of platelet transfusion still require further validation based on large-sample data. In summary, investigating the correlation between platelet transfusion during ICU stay and 28-day mortality in SAT patients, as well as evaluating the impact of platelet transfusion on bleeding, thrombotic events, and inflammation control, is of great significance for optimizing SAT management strategies. This study aims to analyze the effect of platelet transfusion on the prognosis of SAT patients, thereby providing an evidence-based foundation for clinical decision-making.

DETAILED DESCRIPTION:
Sepsis is the most common cause of thrombocytopenia in intensive care unit (ICU) patients, with an incidence rate as high as 35%-59%. Severe thrombocytopenia (≤50×10⁹/L) accounts for 30% of cases, and the degree of thrombocytopenia is positively correlated with mortality risk [1-3]. Studies have shown that patients with sepsis-associated thrombocytopenia (SAT) not only experience prolonged ICU stays and mechanical ventilation duration but also have significantly increased rates of major bleeding events and renal replacement therapy. Meanwhile, the 28-day mortality rate rises with the severity of thrombocytopenia [4, 5]. Platelets play a dual role in sepsis: on one hand, they act as "innocent bystanders" reflecting disease severity; on the other hand, they participate in the pathological process through immune regulation and microvascular protection. For example, platelets contribute to host defense by facilitating neutrophil extracellular traps (NETs) formation mediated by Toll-like receptor 4 (TLR4), but a reduction in platelet count can lead to impaired endothelial barrier function, exacerbating organ edema and bleeding risk [6, 7]. Furthermore, dynamic changes in platelet morphological parameters, such as mean platelet volume (MPV) and platelet distribution width (PDW), are independently associated with inflammatory response and mortality, highlighting the importance of platelet function monitoring [8].

In clinical practice, the primary goal of exogenous platelet transfusion in SAT patients is to rapidly increase circulating platelet counts in cases of inadequate platelet production or excessive consumption, thereby reducing bleeding risk. Due to the complex mechanisms of thrombocytopenia in sepsis-including bone marrow suppression, peripheral consumption (e.g., disseminated intravascular coagulation (DIC), immune-mediated destruction), and splenic sequestration-endogenous platelet recovery is often delayed. Exogenous transfusion provides immediate platelet supplementation, particularly for patients with severe thrombocytopenia (≤50×10⁹/L) accompanied by bleeding tendencies or those requiring invasive procedures (e.g., surgery, central venous catheterization) [9]. Compared to endogenous platelet production (which typically takes 5-7 days), exogenous transfusion helps to rapidly correct hemostatic function, reduce the risk of spontaneous bleeding (such as gastrointestinal or intracranial bleeding); improve endothelial barrier function, decrease microvascular leakage, thereby alleviating organ edema and hypoxic injury; and provide platelets with immunomodulatory activity, potentially regulating excessive inflammatory responses through the release of anti-inflammatory factors (e.g., TGF-β, IL-10) [10, 11].

However, current treatment strategies for SAT remain controversial. Some studies indicate that platelet transfusion may increase in-hospital mortality, particularly in patients with severe thrombocytopenia (≤50×10⁹/L), where transfusion is associated with higher 28-day and 90-day mortality rates, along with risks such as transfusion reactions and alloimmunization [12, 13]. Potential mechanisms include: the inflammatory microenvironment in septic patients may cause rapid activation or destruction of transfused platelets, reducing transfusion efficacy; allogeneic platelets may carry pro-inflammatory mediators (e.g., mitochondrial DNA, high mobility group box 1 (HMGB1)), further exacerbating systemic inflammatory response; and transfusion-related complications, such as transfusion-related acute lung injury (TRALI), transfusion-associated circulatory overload (TACO), and alloimmune reactions, may contribute to adverse clinical outcomes [14, 15]. Additionally, recent studies have found that platelet function may be impaired in septic patients (e.g., increased glycoprotein Ibα (GPIbα) shedding), leading to reduced adhesion and aggregation capacity of transfused platelets and potentially worsening endothelial dysfunction [16].

Previous studies on platelet transfusion and outcomes in SAT patients were all based on database analyses. The results showed that platelet transfusion in septic patients with thrombocytopenia was associated with increased mortality [17, 18]. Currently, there are no multicenter studies on platelet transfusion specifically for SAT patients, and the benefits and risks of platelet transfusion still require further validation based on large-sample data.

In summary, investigating the correlation between platelet transfusion during ICU stay and 28-day mortality in SAT patients, as well as evaluating the impact of platelet transfusion on bleeding and thrombotic events and inflammation control, is of great significance for optimizing SAT management strategies. This study aims to analyze the effect of platelet transfusion on the prognosis of SAT patients, thereby providing an evidence-based foundation for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU between January 2021 and May 2024 and subsequently discharged
* Age ≥ 18 years
* Meeting the Sepsis-3.0 diagnostic criteria
* Platelet count < 100 × 10⁹/L at ICU admission
* ICU length of stay ≥ 48 hours

Exclusion Criteria:

* Active bleeding (e.g., major gastrointestinal bleeding, intracranial hemorrhage) or hematologic malignancies (e.g., leukemia, myelodysplastic syndrome, lymphoma);
* Liver cirrhosis (Child-Pugh class B/C), chronic kidney disease (CKD stage 4-5), or autoimmune diseases (e.g., systemic lupus erythematosus);
* Receipt of chemotherapy, immunosuppressants (e.g., cyclosporine, rituximab), or hematopoietic stem cell/solid organ transplantation within 2 weeks;
* Pregnancy or lactation;
* Pre-existing chronic thrombocytopenia (baseline platelet count <100×10⁹/L for >1 month) or long-term use of antiplatelet/anticoagulant drugs (>2 weeks);
* Significant baseline coagulation dysfunction at ICU admission:Prothrombin time (PT) >1.5 times the upper limit of normal; Activated partial thromboplastin time (APTT) >1.5 times the upper limit of normal; Fibrinogen level <1.0 g/L;
* APACHE II score ≥30 within 24 hours of ICU admission;
* Missing >20% of key data (e.g., daily platelet counts, ICU survival status within 28 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Meeting the Sepsis-3.0 diagnostic criteria and platelet count < 100 × 10⁹/L at ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | Survival status from ICU admission to discharge/transfer from the ICU.
  Survival status from ICU admission to discharge/transfer from the ICU.

SECONDARY OUTCOMES:
Bleeding events | Within 28 days from ICU admission or at the time of ICU transfer/discharge.
  Record newly occurring gastrointestinal bleeding, airway bleeding, epistaxis, oral bleeding, and subcutaneous bleeding within 28 days， based on records from the electronic medical record (EMR) or intensive care unit (ICU) information system
Thrombotic events | Within 28 days from ICU admission or at the time of ICU transfer/discharge.
  Record deep vein thrombosis and pulmonary embolism occurring within 28 days， based on records from the electronic medical record (EMR) or intensive care unit (ICU) information system
ICU length of stay within 28 days | within 28 days after ICU admission
Platelet transfusion therapy-related endpoints | Post-transfusion day 1, 3, 5, and 7
  Record dose-response relationship between platelet transfusion frequency/dosage and ICU mortality;Platelet counts on Day 1, Day 3, Day 5, and Day 7 after platelet transfusion.
Laboratory indicator-related endpoints | Post-transfusion day 1, 3, 5, and 7
  Record the dynamic trajectory of platelet counts (e.g., recovery rate, duration of low values, fluctuation amplitude) based on laboratory results; Trends in platelet morphological parameters (MPV, PDW) and inflammatory markers (IL-6, CRP, PCT).

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital， Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No